CLINICAL TRIAL: NCT03595319
Title: Comparison of Median Alveolar Sevoflurane Concentration for Hypotension Between Young and Elderly Patients: Adaptive Clinical Trial
Brief Title: Median Sevoflurane Concentration for Hypotension Between Young and Elderlypatients: Adaptive Clinical Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brasilia University Hospital (Other)
Responsible Party: Principal Investigator, Gabriel Magalhaes Nunes Guimaraes, Head of Anesthesiology, Brasilia University Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: TccFeliciaVictor2018
Record Dates: First submitted 2018-07-12; First posted 2018-07-23 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Hypotension
Keywords: Hypotension; Sevoflurane; Elderly
MeSH Terms: conditions — Hypotension | interventions — Sevoflurane

STUDY DESIGN:
Intervention Model Description: Adaptive up and down methodology. Anesthesia will be induced using etomidate, rocuronium and remifentanil. After intubation and mechanical ventilation, a high fresh gas flow and variable vaporizer target concentration will be used to stabilize the patient's target end tidal sevoflurane in less than two minutes.
  Each patient's target end tidal sevoflurane is determined by the concentration used in the previous patient of the same group and by the incidence of hypotension. If the previous patient suffered hypotension, next patient's target concentration will drop. If there was no hypotension, next patient's target concentration will rise. The first patient on each group will be 2%. Target end tidal will vary 0.4% until the first crossover, then drop to 0.2% until the second crossover and will vary 0.1% thereafter.
Who Masked: Participant
Masking Description: Participant will not know allocation (sevoflurane concentration) and will be under general anesthesia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young patients (Experimental): Patients between 19 and 40 years-old
  Interventions: Drug: Sevoflurane
- Elder patients (Experimental): Older than 65
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — Inhaled sevoflurane until allocated dose (see adaptive protocol)

SUMMARY:
Two arms: elder group, young group. Dixon's up and down adaptive methodology for ED50. Executed after Anesthesia induction for 10min without touching the patient after starting mechanical ventilation.

DETAILED DESCRIPTION:
This adaptive clinical trial will vary target end tidal sevoflurane by 0.4, then by 0.2 and by 0.1 thereafter in order to minimize sample size.

ELIGIBILITY:
Inclusion Criteria:

* Understands experiment, is voluntary, signs informed consent;
* Does not take medication that influences arterial pressure;
* Normotensive.

Exclusion Criteria:

* Received any medication that influences arterial pressure before experiment;

Ages: 19 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-07-23 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-02-15 (Estimated)

PRIMARY OUTCOMES:
Hypotension incidence related to sevoflurane | During the first 10 minutes after end tidal sevoflurane concentration stabilizes
  Any mean arterial pressure drop > 10% compared to baseline

SECONDARY OUTCOMES:
Systolic hypotension | During the first 10 minutes after end tidal sevoflurane concentration stabilizes
  Systolic arterial pressure drop >10%
Diastolic hypotension | During the first 10 minutes after end tidal sevoflurane concentration stabilizes
  Systolic arterial pressure drop >10%

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel MN Guimarães, MD, MSc, Principal Investigator — University of Brasilia
Locations (1):
- Hospital Universitário de Brasilia, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Plan to share unidentified individual patient data in mendeley data.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Up until mendeley data can host
Access Criteria: Open access
URL: http://www.anestesiologiaunb.com.br